CLINICAL TRIAL: NCT03830593
Title: Is There Anything New in the Field of Large Adrenal Tumors ?
Brief Title: Laparoscopic Adrenalectomy for Large Adrenal Tumors.
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mehmet Necmettin Mercimek, MD, Samsun Liv Hospital
Other Study IDs: OMU KAEK (2019/78)
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2018-12

CONDITIONS: Adrenal Tumor; Adrenal Adenoma
Keywords: endocrine surgery; laparoscopic adrenalectomy;
MeSH Terms: conditions — Adrenal Gland Neoplasms; ACTH Syndrome, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: laparoscopic adrenalectomy group 1: tumor size as < 6 (group1)
  Interventions: Procedure: Laparoscopic Adrenalectomy
- Group 2: Laparoscopic adrenalectomy group2: tumor size ≥ 6 cm (group2)
  Interventions: Procedure: Laparoscopic Adrenalectomy
- Learning Curve: The patients, underwent laparoscopic adrenalectomy, were also classified into group A (1-25), B (26-50), C (51-75), and D (76-102) according to the chronological order of their surgery in order to evaluate the learning curve.
  Interventions: Procedure: Laparoscopic Adrenalectomy

INTERVENTIONS:
Procedure: Laparoscopic Adrenalectomy — minimally invasive lateral transperitoneal adrenalectomy

SUMMARY:
Laparoscopic adrenalectomy is the treatment of choice for the benign tumor of less than 6 cm. However, this is an ongoing debate that exact cut-off value of tumor size for LA. The aim of this study was to assess whether the size of the adrenal tumor affects preoperative and postoperative outcomes in patients undergoing laparoscopic transperitoneal adrenalectomy as well as to evaluate the learning curve.

DETAILED DESCRIPTION:
From April 2010 to October 2018, preoperative and postoperative data of 107 patients who underwent LTA with adrenal mass were recorded prospectively and analyzed retrospectively.

The inclusion criteria were all hormonally active adrenal lesions, detection of increases in size in < 4 cm adrenal tumors on serial imaging, solitary adrenal metastases without evidence of local invasion, tumors size ≥ 4 cm, patients between the age of 18 and 80, and American Society of Anesthesiologists score (ASA) ≤ 3. The patients with adrenal masses that specified suspicion of malignancy on imaging such as local invasion, irregular tumor margins were evaluated as ineligible for LTA, and excluded in this study, were addressed to open surgery. Retroperitoneoscopic and laparoscopic partial adrenalectomies were also excluded from the study.

Totally 102 patients were included in the study. The patients were allocated according to adrenal tumor size as <6cm (group 1:76) and ≥ 6 cm (group 2: 26). The variables such as demographics, tumor size, and laterality, operation time, blood loss, per-operative and postoperative complications, length of hospital stay, final pathology result were compared between the two groups. In order to evaluate the learning curve, the patients were also classified into three consecutive groups including group A (1-25), group B (25-50), group C (51-75) and group D (76-102) according to the chronological order of their surgery. Variables including operation time, tumor size, blood loss, and hospital stay, and overall complications were used to investigate the learning curve.

ELIGIBILITY:
Inclusion Criteria:

1. all hormonally active adrenal lesions,
2. detection of increases in size in < 4 cm adrenal tumors on serial imaging,
3. solitary adrenal metastases without evidence of local invasion,
4. tumors size ≥ 4 cm,
5. patients between the age of 18 and 80
6. American Society of Anesthesiologists score (ASA) ≤ 3.

Exclusion Criteria:

1. suspicion of malignancy on imaging such as local invasion, irregular tumor margins
2. Retroperitoneoscopic adrenalectomies
3. laparoscopic partial adrenalectomies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From April 2010 to October 2018, preoperative and postoperative data of 107 patients who underwent laparoscopic adrenalectomy
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Operation time | intraoperative (minute)
  time from onset to complete of operation
Blood loss | intraoperative
  amount of bleeding during surgery (milliliter)
hospitalization | 1 day
  duration of postoperative hospital stay
Complication | 1 day
  abnormal conditions during or after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Şaban Sarıkaya, Prof. MD, Study Chair — Ondokuz Mayıs University
Locations (2):
- Turkey (Türkiye) (2):
  - Samsun Liv Hospital, Samsun
  - Ondokuz Mayıs University, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huynh KT, Lee DY, Lau BJ, Flaherty DC, Lee J, Goldfarb M. Impact of Laparoscopic Adrenalectomy on Overall Survival in Patients with Nonmetastatic Adrenocortical Carcinoma. J Am Coll Surg. 2016 Sep;223(3):485-92. doi: 10.1016/j.jamcollsurg.2016.05.015. Epub 2016 May 26. PMID 27238874
- [Result] Conzo G, Gambardella C, Candela G, Sanguinetti A, Polistena A, Clarizia G, Patrone R, Di Capua F, Offi C, Musella M, Iorio S, Bellastella G, Pasquali D, De Bellis A, Sinisi A, Avenia N. Single center experience with laparoscopic adrenalectomy on a large clinical series. BMC Surg. 2018 Jan 11;18(1):2. doi: 10.1186/s12893-017-0333-8. PMID 29325527